CLINICAL TRIAL: NCT06426537
Title: A Comparative Study of Colchicine's Role in Reducing Cardiac Fibrosis in Acute Myocardial Infarction Patients: Evaluating Outcomes With Percutaneous Coronary Intervention Versus Without Reperfusion
Brief Title: Colchicine's Efficacy in MI Patients: Comparing PCI and Non-Reperfusion Approaches
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Brawijaya (Other)
Responsible Party: Principal Investigator, Tri Astiawati, Dr. Iskak General Hospital, Tulungagung, East Java, Indonesia, University of Brawijaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 400/235/K.3/302/2020
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: ST-Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Colchicine; Tablets

STUDY DESIGN:
Intervention Model Description: This study investigates the impact of Colchicine on patients with ST-Elevation Myocardial Infarction (STEMI) undergoing different treatment strategies, including percutaneous coronary intervention (PCI) and no revascularization.
Who Masked: Participant
Masking Description: The subjects of this study are patients with ST-Elevation Myocardial Infarction (STEMI) who have undergone Percutaneous Coronary Intervention (PCI) and those without reperfusion. Subject selection was conducted using purposive sampling. Patients who received early PCI without reperfusion were divided into four groups: 1). Early PCI with Colchicine, 2). Early PCI with placebo, 3). STEMI without reperfusion with Colchicine and STEMI without reperfusion with placebo. This approach aims to rigorously evaluate the effects of Colchicine in managing inflammation and cardiac remodeling in STEMI patients, comparing its efficacy against standard placebo treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Colchicine Intervention in STEMI Patients Onset < 12 Hours Undergoing PCI (Active Comparator): Patients receive colchicine according to protocol: Loading dose of 1 mg 1-2 hours before PCI, 0.5 mg colchicine 1 hour after loading, Maintenance dose of 1 x 0.5 mg colchicine for 1 month and OMT
  Interventions: Drug: Colchicine 0.5 MG Oral Tablet
- Placebo in STEMI Patients Onset < 12 Hours Undergoing PCI (Placebo Comparator): Patients receive placebo according to protocol: Placebo administration and OMT
  Interventions: Drug: Colchicine 0.5 MG Oral Tablet
- Colchicine Intervention in STEMI Patients Onset < 12 Hours Not Undergoing Reperfusion (Active Comparator): Patients receive colchicine according to protocol: Loading dose of 1 mg, 0.5 mg colchicine 1 hour after loading, Maintenance dose of 1 x 0.5 mg colchicine for 1 month and OMT
  Interventions: Drug: Colchicine 0.5 MG Oral Tablet
- Placebo in STEMI Patients Onset < 12 Hours Not Undergoing Reperfusion (Placebo Comparator): Patients receive placebo according to protocol: Placebo administration and OMT
  Interventions: Drug: Colchicine 0.5 MG Oral Tablet

INTERVENTIONS:
Drug: Colchicine 0.5 MG Oral Tablet — Oral administration of Colchicine in STEMI patients
  Other Names: Colchicine Tablets; Generic Colchicine; Colchicine Oral Administration

SUMMARY:
This study investigates the effect of Colchicine in preventing heart structure changes following ST-segment elevation myocardial infarction. Through a clinical trial involving patients requiring coronary intervention, we explore how Colchicine can reduce inflammation and fibrosis, two crucial factors influencing heart failure post-heart attack. The outcomes are expected to offer new insights into post-heart attack treatments to prevent heart failure.

DETAILED DESCRIPTION:
This clinical trial, a prospective, focuses on patients with ST-Elevation Myocardial Infarction (STEMI) requiring Percutaneous Coronary Intervention (PCI) within 12 hours of onset. The study aims to control bias effectively through randomization, evenly distributing confounding factors across two groups. Patients, unknown to both researchers and themselves whether receiving Colchicine or a placebo, will undergo reperfusion therapy and optimal medicinal treatment according to the latest guidelines. The study population includes all STEMI patients in three cities in East Java (Jember, Malang, Tulungagung), selected through purposive sampling. The independent variable is Colchicine administration, while dependent variables include ventricular remodeling assessed by Left Ventricular End-Diastolic Volume (LVEDV) via echocardiography, serum levels of caspase-1, TGF-β, NT pro BNP and Galectin-3. All patients receive standard medical treatment pre-PCI, including aspirin and antiplatelet drugs, with post-PCI Optical Medical Treatment (OMT) following the latest guidelines.

The trial is randomized, double-blinded, and placebo-controlled, with participants divided into four groups: early PCI with Colchicine or placebo, and STEMI without reperfusion, receiving either Colchicine or placebo. This setup allows for a comprehensive comparison across different patient management strategies, exploring Colchicine's potential benefits in post-AMI care and its effects on key inflammatory and fibrotic markers.

ELIGIBILITY:
Inclusion Criteria:

Men and women aged 18 years or older. Able and willing to provide informed consent. Presenting with clinical symptoms and supporting examinations indicative of a first-time diagnosis of IMA-EST.

Eligible for treatment according to the IMA-STEMI guidelines, which may include:

Antiplatelet therapy Renin-angiotensin-aldosterone system inhibitors Beta-blockers

Specifically, includes patients who have:

Undergone early PCI. Not received reperfusion therapy. Female patients must commit to avoiding pregnancy during the study. Willing to participate in follow-up via face-to-face or telephone contact.

Exclusion Criteria:

Presence of concurrent diseases such as infections, inflammation, or malignancy.

Diagnosed with gastrointestinal disorders including Crohn's disease, ulcerative colitis, or exhibiting chronic diarrhea.

Recent abnormal laboratory results (within the last 30 days) including:

Hemoglobin below 11.5 g/L Leukocytes below 3.0 x 10^9/L Platelets below 110 x 10^9/L ALT more than three times the upper limit of normal Total bilirubin more than twice the upper limit of normal Creatinine more than twice the upper limit of normal History of liver cirrhosis, acute hepatitis exacerbation, or severe liver disease.

Currently pregnant, breastfeeding, or planning to become pregnant during the study.

History of alcohol abuse. Receiving long-term steroid therapy or using colchicine for other indications. History of hypersensitivity to colchicine. Severe renal failure (eGFR below 30). History of cardiac arrest, ventricular fibrillation, cardiogenic shock, or hemodynamic instability.

Unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
mpact of Colchicine on Ventricular Remodeling in Acute ST-Elevation Myocardial Infarction (STEMI) Patients Post-PCI | Baseline and 1 month post-intervention
  This study assesses the impact of colchicine on ventricular remodeling by measuring changes in the expression of NLRP3 inflammasome, TGF-β, and galectin-3. These biomarkers are indicative of inflammation and fibrotic activity affecting ventricular structure and function in acute STEMI patients post-PCI or without reperfusion therapy

CONTACTS AND LOCATIONS:
Overall Officials: Tri Astiawati, MD. SpJp, Principal Investigator — Dr. Iskak General Hospital, Tulungagung, East Java, Indonesia
Locations (1):
- Tri Astiawati, Tulungagung, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
we will distribute the informed consent form and the study protocol

REFERENCES:
- [Derived] Astiawati T, Rohman MS, Wihastuti T, Sujuti H, Endharti AT, Sargowo D, Oceandy D, Lestari B, Triastuti E, Nugraha RA. Efficacy of Colchicine in Reducing NT-proBNP, Caspase-1, TGF-beta, and Galectin-3 Expression and Improving Echocardiography Parameters in Acute Myocardial Infarction: A Multi-Center, Randomized, Placebo-Controlled, Double-Blinded Clinical Trial. J Clin Med. 2025 Feb 18;14(4):1347. doi: 10.3390/jcm14041347. PMID 40004876
- Available data/document: Study Protocol — http://drive.google.com/drive/u/3/folders/15qW39gHRtgwIuP8rGm8ukhXtYnLRCFNO